CLINICAL TRIAL: NCT02299518
Title: Phase 1 Study of Selinexor in Combination With Topoisomerase-II Inhibition in Acute Myeloid Leukemia
Brief Title: Selinexor and Chemotherapy in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alice Mims (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Alice Mims, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU 14089; NCI-2014-02229 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-11-19; First posted 2014-11-24 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Mitoxantrone; Etoposide; Cytarabine; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (mitoxantrone, etoposide, cytarabine, selinexor) (Experimental): Patients receive mitoxantrone hydrochloride IV, etoposide IV, and cytarabine IV QD on days 1-6 and selinexor PO on days 1, 3, 8, 10, 15, and 17. Treatment continues for 1 course (28 days). Further treatment is based on disease response. Patients achieving CR/CRi are evaluated for stem cell transplant; patients who do not proceed to transplant may receive selinexor as monotherapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: mitoxantrone hydrochloride; Drug: etoposide; Drug: cytarabine; Drug: selinexor; Other: laboratory biomarker analysis; Other: pharmacological study
- Cohort B (etoposide, selinexor) (Experimental): Patients receive etoposide PO QD on days 1-5 and selinexor PO on days 1, 3, 8, 10, 15, and 17. Treatment may repeat every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving response after 4 courses discontinue treatment; patients achieving response may receive up to 4 courses of maintenance therapy every 8 weeks. Patients may then continue selinexor as monotherapy at the discretion of the principal investigator.
  Interventions: Drug: etoposide; Drug: selinexor; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ
  Arms: Cohort A (mitoxantrone, etoposide, cytarabine, selinexor)
Drug: etoposide — Given IV and PO
  Other Names: EPEG; VP-16; VP-16-213
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
  Arms: Cohort A (mitoxantrone, etoposide, cytarabine, selinexor)
Drug: selinexor — Given PO
  Other Names: CRM1 nuclear export inhibitor KPT-330; KPT-330; selective inhibitor of nuclear export KPT-330; SINE KPT-330
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of selinexor when given together with etoposide with or without mitoxantrone hydrochloride and cytarabine in treating patients with acute myeloid leukemia that has returned (relapsed) or has not responded to treatment (refractory). Selinexor may help stop the growth of tumor cells by blocking an enzyme needed for cancer cell growth. Drugs used in chemotherapy, such as etoposide, mitoxantrone hydrochloride, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy together with selinexor work better in treating relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of selinexor in combination with mitoxantrone hydrochloride, etoposide, cytarabine (MEC) or oral etoposide (respective cohorts are independent of each other) in patients with relapsed or refractory acute myeloid leukemia (AML).

II. To define the specific toxicities, maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of these combinations.

III. To determine the recommended phase 2 dose (RP2D) of these combinations.

SECONDARY OBJECTIVES:

I. To determine the rate and duration of complete remission (CR) ± hematologic recovery of selinexor plus MEC therapy in AML.

II. To determine the overall response rate (ORR). III. To define the rate of complete remission (CR + CR with incomplete blood count recovery [CRi]) rate by the end of induction therapy.

IV. Determine the disease-free survival for patients who reached CR/CRi within 1 year.

TERTIARY OBJECTIVES:

I. To conduct pharmacodynamic studies by measuring the effect of these chemotherapy combinations on the inhibition of exportin 1 (XPO1).

II. To conduct pharmacokinetic sampling of selinexor and etoposide at limited time points to assess drug metabolism, peak plasma levels and area under curve (AUC).

OUTLINE: This is a dose-escalation study of selinexor. Patients are assigned to 1 of 2 cohorts.

COHORT A (PATIENTS FIT FOR INTENSIVE THERAPY, AGE < 60): Patients receive mitoxantrone hydrochloride intravenously (IV), etoposide IV, and cytarabine IV once daily (QD) on days 1-6 and selinexor orally (PO) on days 1, 3, 8, 10, 15, and 17. Treatment continues for 1 course (28 days). Further treatment is based on disease response. Patients achieving CR/CRi are evaluated for stem cell transplant; patients who do not proceed to transplant may receive selinexor as monotherapy in the absence of disease progression or unacceptable toxicity.

COHORT B (PATIENTS UNFIT FOR INTENSIVE THERAPY, AGE ≥ 60): Patients receive etoposide PO QD on days 1-5 and selinexor PO on days 1, 3, 8, 10, 15, and 17. Treatment may repeat every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients not achieving response after 4 courses discontinue treatment; patients achieving response may receive up to 4 courses of maintenance therapy every 8 weeks. Patients may then continue selinexor as monotherapy at the discretion of the principal investigator.

After completion of study treatment, patients are followed up for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory AML; Cohort A patients must be < 60 years of age and have failed at least one prior induction regimen for AML; Cohort B patients must be ≥ 60 years of age, unfit for intensive therapy (physician opinion), and have failed an induction regimen for AML. The maximum number of prior lines of induction for both cohorts is 3
* Patients with secondary AML or therapy related disease (t-AML) are eligible
* If the patient has co-morbid medical illness, life expectancy attributed to this must be greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin < 2.0 mg/dL, except when patient is known to have Gilbert's Syndrome, the total bilirubin can be ≤3.0 mg/dL.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal
* Creatinine (Cr) clearance > 50 mL/min by Modification of Diet in Renal Disease (MDRD) calculation
* New York Heart Association (NYHA) congestive heart failure (CHF) class II or better
* Cardiac ejection fraction >= 50%
* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential; acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal; for both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose
* Ability to understand and willingness to sign the written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients receiving any other investigational agents or patients that have received other investigational agents within 14 days of enrollment
* Patients with active central nervous system (CNS) malignancy; asymptomatic small lesions are not considered active; treated lesions may be considered inactive if they are stable for at least 3 months; patients with malignant cells in their cerebrospinal fluid (CSF) without CNS symptoms may be included
* Major surgery within 2 weeks before day 1
* Uncontrolled active infection; patients with infection requiring parenteral antibiotics are eligible if the infection is controlled
* Patients with significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea
* History of seizures, movement disorders or cerebrovascular accident within the past 3 years prior to cycle 1 day 1
* Patients with macular degeneration, uncontrolled glaucoma, or markedly decreased visual acuity
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association [NYHA) class III or IV), unstable angina pectoris, myocardial infarction within 6 months prior to enrollment, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Pregnant women or women who are breastfeeding are excluded from this study; confirmation that the subject is not pregnant must be established by a negative serum beta (β)-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patients with advanced malignant solid tumors
* Patients whom, in the opinion of the investigators, are significantly below their ideal body weight
* Patients who are not able to swallow capsules or tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
MTD of selinexor, defined as the highest safely tolerated dose where, at most, one patient experiences DLT in 6 evaluable patients, with the next higher dose having at least 2 patients who experience DLT | 28 days
  The National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 will be used to characterize toxicities.

SECONDARY OUTCOMES:
Degree of response | Up to 30 days after completion of study treatment
  Summarized within each stratum and at each dose level.
Duration of response | Up to 30 days after completion of study treatment
  Duration of response will be reported for patients who achieve complete remission.
ORR | Up to 30 days after completion of study treatment
  Will be presented for those patients treated at the MTD with an exact 95% confidence interval.

OTHER OUTCOMES:
Change in expression of XPO1 and surrogates or direct targets of XPO1 | Baseline to up to day 35 (Cohort A) or day 29 of last course of treatment (Cohort B)
  The impact of selinexor on the inhibition of XPO1 expression and various genes/microribonucleic acids that serve as surrogates or direct targets of XPO1 will be characterized. Expression prior to administration of selinexor and following treatment with selinexor will be described graphically using boxplots or summary measures (e.g. mean and standard errors). Trends of dose response will be explored within each stratum, as well as whether targets are being "hit" between the strata. Due to data limitations in early clinical trials, analyses will be descriptive in nature.
Plasma pharmacokinetic (PK) parameters of selinexor will be assessed for oral and IV using non-compartmental and compartmental methods. | 1, 2, 4 and 24 hours post-dose days 1 and 15 of course 1; pre-dose days 3 and 17 of course 1
  Intracellular PK of selinexor will be evaluated primarily by determining total intracellular concentrations of parent drugs on day 1 and day 8. The primary hypothesis is that selinexor intracellular exposure (area under the concentration-time curve, AUCIC), normalized to plasma exposure (AUCP), will be greater on Day 1 vs. Day 8 due to reduced intracellular selinexor-glutathione conjugation in the presence of etoposide. The AUCIC and AUCIC/AUCP ratio will be evaluated for correlations with selinexor activity."
Plasma pharmacokinetic (PK) parameters of etoposide and will be assessed for oral and IV using non-compartmental and compartmental methods. | 1, 2, 4 and 24 hours post-dose days 1 and 15 of course 1; pre-dose days 3 and 17 of course 1
  Intracellular PK of etoposide will be evaluated primarily by determining total intracellular concentrations of parent drugs on day 1 and day 8. The primary hypothesis is that selinexor intracellular exposure (area under the concentration-time curve, AUCIC), normalized to plasma exposure (AUCP), will be greater on Day 1 vs. Day 8 due to reduced intracellular selinexor-glutathione conjugation in the presence of etoposide. The AUCIC and AUCIC/AUCP ratio will be evaluated for correlations with selinexor activity."

CONTACTS AND LOCATIONS:
Overall Officials: Alice Mims, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- The State Ohio University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Bhatnagar B, Zhao Q, Mims AS, Vasu S, Behbehani GK, Larkin K, Blachly JS, Badawi MA, Hill KL, Dzwigalski KR, Phelps MA, Blum W, Klisovic RB, Ruppert AS, Ranganathan P, Walker AR, Garzon R. Phase 1 study of selinexor in combination with salvage chemotherapy in Adults with relapsed or refractory Acute myeloid leukemia. Leuk Lymphoma. 2023 Dec;64(13):2091-2100. doi: 10.1080/10428194.2023.2253480. Epub 2023 Sep 4. PMID 37665178
- See also: The Jamesline — http://cancer.osu.edu